CLINICAL TRIAL: NCT01149161
Title: Sentinel Lymph Node Biopsy in the Thyroid Carcinoma; Randomized, Prospective Study
Brief Title: Extent of Central Lymph Node Dissection in Papillary Thyroid Microcarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jee soo Kim, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-02-017
Record Dates: First submitted 2010-06-02; First posted 2010-06-23 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma
Keywords: neck dissection; sentinel lymph node; Carcinoma; Papillary; thyroid; dissection
MeSH Terms: conditions — Carcinoma; Thyroid Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C group (Active Comparator): Routine central neck dissection
  Interventions: Procedure: Routine central neck dissection
- N group (No Intervention): No central neck node dissection

INTERVENTIONS:
Procedure: Routine central neck dissection — Level VI neck node dissection during thyroid operation
  Arms: C group

SUMMARY:
Occult lymph node metastasis is common in micro papillary thyroid cancer. However, the role of lymph node dissection in the treatment of microPTC remains controversial. The investigators want to investigate the usefulness routine central dissection and sentinel lymph node biopsy in prognosis of micro PTC. This is a prospective randomized control study. The investigators started this study from May of 2009 and this study will be continued until Dec. 2011.

DETAILED DESCRIPTION:
The investigators will assign all patients to three groups; no dissection group (Group I), sentinel lymph node biopsy only group (Group II) and routine central neck dissection group (Group III). At first, to know the necessity of routine central neck node dissection for micro PTC,the investigators will compare the result of group I and group III. Additionally, the investigators can analyze the usefulness of sentinel lymph node biopsy for substitution of routine central neck node dissection for micro PTC.

ELIGIBILITY:
Inclusion Criteria:

* papillary carcinoma of thyroid (less than 4cm)
* no evidence of lymph node metastasis in preoperative work-up result
* the patients who accept this study

Exclusion Criteria:

* large thyroid cancer( > 4cm)
* morbid
* anticoagulation agent usage
* endoscopic or robotic thyroid operation
* evidence of lymph node metastasis or extrathyroidal extension in preoperative US and CT scan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2009-05; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Is routine neck node dissection necessary in micro PTC? | Until 5 year follow-up. (Dec. 2016)
  To see the necessity of routine neck node dissection in micro PTC, we will compare the recurrence rate and other complication (e.g. hoarseness and hypocalcemia) between group I(no dissection) and group III(routine dissection) after completion of study(after 5 year f/u).
  To check the safety of this study, our result will be checked by korea institutional reveiw board every one year.

SECONDARY OUTCOMES:
The efficacy of sentinel lymph node biopsy in micro PTC | Until 5 year follow-up. (Dec. 2016)

CONTACTS AND LOCATIONS:
Overall Officials: Jee Soo Kim, M.D., Ph.D., Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No